CLINICAL TRIAL: NCT02622503
Title: Retrospective Data Collection on Rheumatoid Arthritis (RA) Patients Treated With Rituximab in Finland.
Brief Title: A Study on Rheumatoid Arthritis Patients Treated With Rituximab
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30146
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis: Patients with rheumatoid arthritis receiving rituximab will be observed for treatment responses.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — This is an observational study. Patients with rheumatoid arthritis and having received treatment previously will be assessed for the treatment responses.

SUMMARY:
The purpose of the study is to obtain an overall picture of rituximab treatments and treatment responses in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA) patients treated with rituximab in Finland

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatoid arthritis (RA) patients treated with rituximab in Finland.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Information on previous RA treatments | 3 months
Information on rituximab treatment responses | 3 months
Information on concomitant medications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Finland (5):
  - Helsinki
  - Jyväskylä
  - Lahti
  - Tampere
  - Turku